CLINICAL TRIAL: NCT06702553
Title: Effect of Inhaled Nitric Oxide on Major Adverse Events Requiring Intensive Life Support in Adults Undergoing Cardiac Surgery With Cardiopulmonary Bypass: A Phase III, Double-Blind, Multicenter, Randomized Controlled Trial (Nitric Oxide for Reduced Intensive Support in Cardiac Surgery With Cardiopulmonary Bypass, the NORISC Trial)
Brief Title: Nitric Oxide for Reduced Intensive Support in Cardiac Surgery With Cardiopulmonary Bypass
Acronym: NORISC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Collaborators: Nikolay O. Kamenshchikov., M.D., Tomsk National Research Medical Center of the Russian Academy of Sciences (Unknown); Lorenzo Berra., M.D., Massachusetts General Hospital (Unknown); Jiange Han, Tianjin Chest Hospital, Tianjin, China (Unknown); Qingping Wu, Wuhan Union Hospital, Wuhan, China (Unknown); Evgeniy Grigoriev, Research Institute for Complex Issues of Cardiovascular Diseases, Kemerovo, Russian Federation (Unknown); Vladimir Boboshko, E. Meshalkin National Medical Research Center, Novosibirsk, Russian Federation (Unknown); Andrei Bautin, The Almazov National Medical Research Centre, St. Petersburg, Russian Federation (Unknown); Vladimir Pichugin, Specialized Cardiac Surgery Clinical Hospital named after Academician B.A. Korolev, Nizhny Novgorod, Russian Federation (Unknown); Evgeniy Rosseykin, Federal Center of Cardiovascular Surgery, Khabarovsk, Russian Federation (Unknown); Sheng Wang, Anzhen Hospital, Beijing, China (Unknown)
Responsible Party: Principal Investigator, Chong Lei, MD & phD, Principal Investigator, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY20242322
Record Dates: First submitted 2024-11-18; First posted 2024-11-25 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-04

CONDITIONS: Nitric Oxide; Cardiac Surgery; Cardiopulmonary Bypass; Adult Patients Undergoing Cardiovascular Surgery With Cardiopulmonary Bypass
Keywords: Nitric Oxide; cardiopulmonary bypass; major adverse events; cardiac surgery; complications; Organ protection
MeSH Terms: interventions — Endothelium-Dependent Relaxing Factors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The intervention gas tanks and the gas delivery systems or the intervention gas generator system in the OR and at the bedside when patients in ICU are covered with drapes and masked that cannot be distinguished on the basis of appearance. This allows to keep participants, clinicians and investigators blind to the assignment group. For safety and gas monitoring, the clinician (or respiratory therapist) administering the test gas remains unblinded to the treatment. This unblinded clinician(or respiratory therapist) is solely responsible for gas tank preparation and test gas delivery and monitoring.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention: iNO Group (Experimental): Patients will receive 80 parts per million (ppm) NO during CPB through the oxygenator. After weaning of CPB, test gases will be delivered via inspiration limb of ventilator at a dose range of 40-80 ppm until 6 hours after ICU admission or until extubation after surgery, whichever comes first.
  Interventions: Drug: Nitric Oxide Gas
- Standard Care/Control Group (Placebo Comparator): Patients in this group will receive standard care and 80 ppm nitrogen (N2, control group) are added to the gas mixture as control. In the circumstances when the N2 is not applicable, such as when the plasma-chemical NO synthesis device is employed for NO generatiaon and delivery, the device will be connected to the CPB and ventilator circuits, but the synthesis will remain inactive in the control group. Consequently, the circuit will be supplied with air devoid of NO.
  Interventions: Drug: Standard Care Arm

INTERVENTIONS:
Drug: Nitric Oxide Gas — Patients will receive 80 parts per million (ppm) NO during CPB through the oxygenator. After weaning of CPB, test gases will be delivered via inspiration limb of ventilator at a dose range of 40-80 ppm until 6 hours after ICU admission or until extubation after surgery, whichever comes first.
  Other Names: Nitric Oxide inhalation
  Arms: Intervention: iNO Group
Drug: Standard Care Arm — Patients in this group will receive standard care and 80 ppm nitrogen (N2, control group) are added to the gas mixture as control. In the circumstances when the N2 is not applicable, such as when the plasma-chemical NO synthesis device is employed for NO generatiaon and delivery, the device will be connected to the CPB and ventilator circuits, but the synthesis will remain inactive in the control group. Consequently, the circuit will be supplied with air devoid of NO.
  Other Names: Nitrogen inhalation
  Arms: Standard Care/Control Group

SUMMARY:
Cardiac surgery is a procedure that is commonly performed worldwide. Despite these technological advances, cardiac surgery remains a high-risk surgery. Among post-operative complications, acute kidney injury, respiratory failure, myocardial infarction, and stroke as well as cognitive dysfunction are significant causes of mortality in patients undergoing and following cardiac surgery. Inhaled nitric oxide (NO) therapy as a selective pulmonary vasodilator in cardiac surgery has been one of the most significant pharmacological advances in managing pulmonary hemodynamics and life threatening right ventricular dysfunction and failure. In addition, newer applications show greater promise of inhaled NO as a therapy in the area of cardiac surgery associated acute kidney injury and ischemia reperfusion. However, this remarkable expectation to inhaled NO has experienced a roller-coaster ride with high hopes and nearly universal demonstration of physiological benefits but disappointing translation of these benefits to harder clinical outcomes, like mortality. Most of our understanding on the iNO field in cardiac surgery stems from small observational or single center randomized trials, which failed to ascertain strong evidence base. As a consequence, there are only week clinical practice guidelines on the field and only European expert opinion for the use of iNO in routine and more specialized cardiac surgery. There is need for a large multicenter randomized controlled study to confirm the administration of iNO as an effective weapon for the battle against life threatening complication in high risk cardiac surgical patients.

In a previous meta analysis with 27 studies included, we demonstrated that inhaled nitric oxide (NO) could reduce the duration of mechanical ventilation and reducing biomarkers of organ injury and clinical signs of organ dysfunction in cardiac surgery under cardiopulmonary bypass (CPB) , but had no significance in the ICU stay, hospital stay, and mortality. This may be attributed to the small sample size of the most included studies (of the 27 studies included, 20 studies with sample size less than 100) and heterogeneity in timing, dosage and duration of iNO administration. Well-designed, large-scale, multicenter clinical trials are needed to further explore the effect of iNO in improving postoperative prognosis in cardiovascular surgical patients.

We are planning a large multicenter controlled randomized trial to demonstrate that inhaled nitric oxide can reduce composite outcome of death and Major Adverse Events (MAEs), including need for intensive supports due to heart failure, low cardiac output sydrome, or renal failure, respiratory failure, etc., and myocardial infarction, stroke, and sepsis at 30 days after surgery from 20% to 16% in patient undergoing cardiac surgery with cardiopulmonary bypass.

If the hypothesis had been proved and validated, the results of this study can provide strong evidence for guidelines to facilitate the routine use of iNO in all cardiopulmonary bypass assisted cardiac procedures with 31,800 postoperative outcomes improved per year in US and in China.

DETAILED DESCRIPTION:
Cardiac surgery is a procedure that is commonly performed worldwide, and often requires the use of the cardiopulmonary bypass (CPB) machine to perform surgery on a non-beating heart. It was reported that the total volume of all cardiac surgical procedures in 2019 was 301,077 in US7 and 263, 292 in China in 2022, respectively.

Diseases of cardiovascular system confidently occupy the first place among the causes of disability and mortality in developed countries. In recent years, many clinicians, scientists, and engineers have been involved in efforts to develop safer procedures, novel biomaterials, heart substitutes, life-support systems, and safer methods to control cardiac arrhythmias and improve ventricular remodeling after injury. Progress in medicine over the past decades is clearly manifested in the rapid development of cardiovascular surgery. Despite these technological advances, cardiac surgery remains a high-risk surgery.

Cardiac surgery is accompanied by a number of complications. The perioperative mortality rate in the general population of cardiac surgery patients ranges from 2 to 10% depending on the type of surgery, the severity of left ventricular dysfunction and the presence of concomitant diseases . This pattern is true even for routine interventions with a relatively low risk of organ dysfunction , and with certain types of operations (combined interventions, reconstructive interventions on the ascending aorta and aortic arch, multivalve heart surgery) the incidence of severe organ dysfunction can increase to 70% with the need for supportive therapy in 16% of cases. Fundamental rationale, development and implementation of perioperative organ protection technologies into clinical practice will save the lives of up to 20 thousand people a year and save up to 1 billion US dollars for the healthcare system.

The search for an optimal strategy for adjuvant organ protection continues. It is extremely promising to identify potential pharmacological agents that are direct triggers or mediators of the implementation of the organoprotective phenotype during cardiac surgery. Among post-operative complications, acute kidney injury and renal failure, prolonged ventilation, myocardial infarction, and stroke as well as cognitive dysfunction are significant causes of mortality in patients undergoing and following cardiac surgery.

Inhaled nitric oxide (NO) is a selective pulmonary vasodilator approved by the U.S. Food and Drug Administration(FDA) in 1999 for the treatment of persistent pulmonary hypertension of the newborn(PPHN). Inhaled NO has been largely used in Europe since 1992, and obtained the status of drug in France in 2001 and in Belgium in 2008. The European market authorizations (MA) defined 2 labeled indications: PPHN and treatment of PH related to cardiac surgery. The most common scenario for the commencement of iNO therapy in rountine cardiac surgery is postoperative right ventricular dysfunction of failure in the setting of increased pulmonary vascular resistance, which is related to pulmonary hypo-perfusion or activation of systemic inflammatory response. Cardiac procedures with prolonged CPB are associated with progressively high level of hemolysis, causing the release of free hemoglobin (fHb) and increase of NO inhibitor asymmetric dimethylarginine. The deoxygenation reaction with fHb and the inhibition of the endothelial NO synthetase cause vascular NO depletion leading to endothelial dysfunction and vasoconstriction. Inhaling NO can oxidize plasma Oxy-Hb to Met-Hb, thereby reducing plasma NO scavenging in the context of hemolysis. In a previous study, iNO showed promising benefits in lowering plasma NO consumption in presence of hemolysis. Supplementing NO into the CPB circuit could reduce NO consumption, possibly lowering postoperative systemic and pulmonary vascular resistance, and thus improving ventriculo-arterial coupling, cardiac output, and organ perfusion. In addition, CPB could induce systemic inflammation due to ischemic-reperfusion injury, which could contribute to myocardial dysfunction and to further decrease endogenous NO production. In this setting, inhaled NO could exert immune modulation and limit myocardial dysfunction. As many aspects of cardiac surgery including the pulmonary ischemia, the deleterious effects of cardiopulmonary bypass on pulmonary vasoactive impacts on PVR, endothelial dysfunction and NO pathways, treatment by supplemental delivery of NO seems logical. iNO has also been used following cardiac surgery, including after heart transplant to reduce afterload on the right ventricle with the goal of augmenting cardiac output and decreasing the risk of RV failure.

Two studies have been released showing that the addition of gaseous NO into the CPB circuit resulted in myocardial protection, a reduction in the length of mechanical ventilation, and postulated that this effect may be due to the anti-inflammatory properties of NO.In a recent multicenter, double-blind, randomized controlled trial of inhalation of NO in 250 patients with ST-elevation myocardial infarction (STEMI). Inhalation of NO at 80 ppm for 4 hrs in these patients after cardiac catheterization was safe, and there was a tendency toward decreased rates of adverse events at 4 months (P=0.10) and 1 year (P=0.06) in patients who received NO. The improvement in cardiac output in response to inhaled NO in patient undergoing cardiac surgery had been demonstrated in series of studies, the existing evidence fails to provide long-term morbidity or mortality data to support a benefit of these agents on clinical outcomes. Based on the available clinical evidence, there are only weak clinical practice guidelines on the field and only European expert opinion for the use of iNO in routine and more specialized cardiac surgery. There is need for a large multicenter randomized controlled study to confirm the administration of iNO as an effective weapon for the battle against life threatening complication in high risk cardiac surgical patients.

The improvement in cardiac output in response to inhaled NO in patient undergoing cardiac surgery had been demonstrated in series of studies, the existing evidence fails to provide long-term morbidity or mortality data to support a benefit of these agents on clinical outcomes. Recent evidence continued to demonstrate biological benefits, hemodynamically important physiological benefit and have begun to demonstrate some meaningful clinical outcomes such as reduction in duration of mechanical ventilation and stay in the intensive care unit. A few isolated reports also have suggested that the administration of inhaled NO improved the ability to separate from cardiopulmonary bypass during cardiac operations, decreased the need for inotropic or vasopressor support, decreased the duration of postoperative mechanical ventilation, and decreased intensive care unit (ICU) length of stay. It was demonstrated that iNO led to a small reduction of ICU stay in patients undergoing valve surgery in a sub analysis of a systemic review of 18 RCTs of adult cardiac surgery. However, these observed benefits have not been reproduced in other studies.

Whether or not treatment of pulmonary hypertension with Inhaled NO during cardiac surgery alters clinically important patient outcomes (ie, mortality and the length of ICU stay and hospitalization) is unknown. Recent systemic review that NO has minimal or null effect on major clinical outcomes. In a recent systemic review and meta-analysis of 10 studies including 434 patients, The authors concluded that inhaled NO improved right ventricular performance when compared to intravenously administered agents. However, iNO were not superior to placebo in terms of decreasing mortality and had no effect on length of hospitalization in adult patients undergoing cardiac surgery with cardiopulmonary bypass. The therapeutic potential of NO, combined with a good safety profile, justifies its use, despite the lack of definitive evidence demonstrating improved long-term outcomes or survival among cardiac surgery patients, heart transplant patients, lung transplant patients, and patients with implantable mechanical circulatory support devices. Despite an almost 30-year history of use, there is still no convincing evidence base and clear recommendations for the use of NO in cardiac surgery. There is insufficient evidence to reach a consensus regarding dosage, duration of therapy, or effect on patient outcomes, even for routine indications.

Based on the available clinical evidence, there are only weak clinical practice guidelines on the field and only European expert opinion for the use of iNO in routine and more specialized cardiac surgery. There is need for a large multicenter randomized controlled study to confirm the administration of iNO as an effective weapon for the battle against life threatening complication in high risk cardiac surgical patients.

Of the complications, acute kidney injury (AKI) is the single most common organ failure associated with cardiac surgery. Epidemiological data report that AKI associated with cardiac surgery may occur in about 30-70% of cases after cardiac surgery requiring CPB and up to 20% of patients need post-operative renal replacement therapy. Occurrence of AKI is associated with prolonged intensive care and step-down unit admission, increased perioperative cost of care, and most significantly, a higher postoperative morbidity and mortality. Prolonged CPB causes hemolysis with high levels of circulating plasma hemoglobin that scavenges NO via the deoxygenation reaction, depleting endogenous NO and casuing vasoconstriction, proximal renal tubular injury, and AKI.

Previously, our research group hypothesized that administration of 80 ppm NO during the prolonged CPB process and thereafter would preserve kidney function by converting plasma Hb into Met-Hb and preventing intrarenal oxidative reactions and NO scavenging. Then we conducted a single center, prospective, randomized, double-blind controlled trial involving 244 patients with normal kidney function who underwent elective multiple valve replacement surgery that required prolonged CPB. Inhaled NO at 80 ppm was delivered at the onset of CPB via the oxygenator and subsequently through the mechanical ventilator for up to 24 hours. The incidence of AKI in patients treated with NO decreased from 64% to 50% (P=0.014). The beneficial impact of NO was associated with a 22% relative risk reduction in AKI incidence, which translated into a 42% relative reduction of chronic renal function impairment. NO treatment resulted in fewer patients transitioning to stage 3 chronic kidney diseases (estimated glomerular filtration rate, eGFR < 60 ml/min/1.73 m2, 18% versus 31%). The Major Adverse Kidney Event (MAKE) index, defined as a composite outcome of loss of 25% of eGFR from baseline, end-stage renal disease requiring a continuous renal replacement therapy, and mortality, at 30 days, 90 days, and 1 year was more than halved in the NO treatment group. Among these Chinese patients requiring prolonged CPB, 80 ppm NO exposure not only decreased AKI incidence, and further reduced the transition to stage 3 CKD at 90 days and 1 year. However, due to the small sample size, only a trend of decreased mortality in the NO group was observed. Furthur, the leading PI of current trial of Russia, Kamenshchikov N.O et al. showed the nephroprotective effect of nitric oxide, by reducing markers of damage and improving the functional status of kidneys in the perioperative period in cardiac surgical patients operated on under CPB. The authors assessed the concentration of pro-inflammatory and anti-inflammatory mediators, the level of plasma free hemoglobin (fHb), as well as hemodynamic parameters, which did not differ significantly between groups. There were no clinically significant increases in NO2 in the inhaled air-gas mixture or serum methemoglobin (MetHb) concentrations.

To date, data from meta-analyses on the effect of nitric oxide on outcomes in cardiac surgery remain contradictory. Thus, it was shown that perioperative delivery of inhaled nitric oxide resulted in no or minimal benefit in patients with pulmonary hypertension undergoing cardiac surgery. In another meta-analysis, 5 studies and 579 patients were enrolled to investigate the effect of NO on renal function in patients undergoing cardiopulmonary bypass. It turned out that NO was associated with reduced risk of AKI when started from the beginning of CPB, which indicates the benefits of NO can only be exerted when NO was administered before the damage caused by CPB occur. The limitation of these systemic review is that the effect of iNO on mortality was not stated. The most recent meta-analysis to date has shown that using inhaled nitric oxide during cardiopulmonary bypass reduces the length of stay in the intensive care unit, and for children, it reduces the duration of mechanical ventilation. Thus, large randomized studies are required to ascertain the effect of NO on clinical outcomes in cardiac surgery under CPB and further determine the dosage, timing and duration of NO administration. A recent updated meta-analysis conducted by the our research group with 27 studies included, the pooled result demonstrated that iNO reduced the duration of mechanical ventilation, no significant benefits were detected on the ICU stay, hospital stay, and mortality in patients undergoing cardiac surgery. This may be attributed to the small sample size of the most included studies and heterogeneity in timing, dosage and duration of iNO administration.

Preliminary data support the effect of inhaled NO on reducing biomarkers of organ injury and clinical signs of organ dysfunction in cardiac surgery under CPB. Potentially, NO may improve clinical outcomes in cardiac surgery. However, the optimal therapeutic regimen for perioperative NO therapy is unknown. For this study, we chose NO concentration doses of up to 40 ppm during mechanical ventilation and 80 ppm during CPB as optimal for maximizing the organ-protective effects, as shown in previous studies, and at the same time such doses are considered safe. The results of current meta-analyses indicate that the strategy of iNO-mediated protection can reduce major complications. We hypothesize that the use of inhaled NO during surgery, during CPB, and also in the early postoperative period in the ICU at concentrations acceptable in clinical practice can prevent major organ failure and reduce the need for intensive replacement/maintenance therapy. The results of this study, if our hypothesis is confirmed, may bring benefits to society as improved outcomes of cardiac surgery, reduction of the financial burden and logistics challenges for the treatment of postoperative complications and subsequent rehabilitation of patients for the healthcare system, as well as the emotional and financial burden on patients and their families. To test this hypothesis we have designed this multicenter RCT.

In this, multi-center, randomized (1:1) controlled, parallel-arm superiority trial, we hypothesized that administration of NO gas starting from the initiation of CPB lasted until 6-hours after ICU admission or until extubation, whichever comes first, will decrease the incidence of major adverse events with reduced needs for intensive life supports, and so as to improved postoperative prognosis. This study was designed to determine whether NO administered during and after cardiac surgery reduces prespecified composite outcomes at 30 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Elective cardiac or aortic surgery requiring CPB
3. Without history of previous open heart surgery.

Exclusion Criteria:

1. Immediate emergency cardiac surgery;
2. Cardiac surgery that requires deep hypothermic circulatory arrest;
3. Planned cardiac surgery for congenital heart disease repair;
4. Planned for heart transplatation
5. Ongoing heart failure or low output syndrome already on intensive support (IABP, ECMO, left ventricular assist device such as impella, mechanical ventilation), left ventricular ejection fraction of < 30% or comparable, equivalent preoperative conditions
6. Already accepted or currently on inhaled NO therapy or inhaled/aerosolized prostacyclin in the week prior to the enrollment;
7. Endstage kidney disease with estimated glomerular filtration rate (eGFR) < 15 ml/min or already on renal replacement surgery.
8. Hemophilia A or B
9. Other terminal stage of chronic disease with life expectancy less than 1 year per evaluation and adjudication of the attending physicians.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3650 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Composite outcome of death and major adverse events requiring intensive life supports | within 30 days after operation
  It is composite outcome including:
  * all cause mortality;
  * ischemic events(myocardial infarction, ischemic stroke, and pulmonary embolism) ,
  * Cardiac arrest that had been successfully resuscitated or new onset of acute cardiac failure (low output syndrome) requiring IABP, ECMO, left ventricular assist device, cardiac dysfunction need for large dose of inotrope support,
    ---Stage 3 AKI or Renal failure that required renal replacement therapy,
  * prolonged mechanical ventilation (> 24h ),
  * re-sternotomy for any indication,
  * major arrhythmia ((Ventricular fibrilliation or ventricular tachycardia after weaning-off cardiopulmonary bypass, new onset atrial fibrillation requiring anticoagulant therapy or other intervention upon discharge from the hospital);
  * sepsis

SECONDARY OUTCOMES:
Total number of major adverse events (MAEs) | within 30 days after operation
  Total number of major adverse events( MAEs) listed as the components of the primary outcomes.
Incidence of the MAEs | within 30 days after operation
  Incidence of the MAEs listed as the components of the primary outcomes.
All AKI incidence | within 7 days of surgery
  AKI incidence which will be diagnosed by KDIGO criteria
Length of mechanical ventilation | within 30 days after operation
  Length of mechanical ventilation in hours
Readmission | within 30 days after operation
  Readmission after hospital discharge
Length of ICU stay | From the date of surgery until the date patient discharge from hospital, assessed up to 1 year
  Length of postoperative ICU stay
Length of postprocedural hospital stays | From the date of surgery until the date patient discharge from hospital, assessed up to 1 year.
  Length of postprocedural hospital stays
All cause 90 d mortality | within 90 days after operation
  Death within 90 days after surgery for any reason
All cause 1 year mortality | within 1 year after operation
  Death within 1 year after surgery.
Change in organ-specific and total sepsis-related SOFA scores | from the day of surgery to postoperative day 7.
  Change in organ-specific and total sepsis-related Sequential Organ Failure Assessment (SOFA) scores from enrollment through study day 7.
Basal level of hemolysis | after entering operation room and before anaesthesia induction
  Serum free hemoglobin levels at baseline (g/L)
Incidence of acute intraoperative hemolysis | Immediately after the end of cardiopulmonary bypass (CPB)
  measurement will be defined based on the level of free hemoglobin after CPB.
The extent of hemolysis progression | taken at immediately after CPB finishes
  Measured based on the free hemoglobin levels at baseline and immediately after CPB (free hemoglobin levels immediately after CPB/ baseline free hemoglobin)

OTHER OUTCOMES:
Blood transfusion | during postoperative hospitalization, with an average of 10 days
  Amount of each type of blood product transfused (red blood cells, fresh frozen plasma, platelets)
Blood loss | during the first 72 hours after surgery
  Total amount of blood loss (chest tube drainage) in ml
Incidence of prolonged cardiovascular support | during postoperative hospitalization, with an average of 10 days.
  cardiovascular support by using inotropes for more than 48 hours
Maximum vasoactive-inotropic score (VIS) | record the maximun of the day for the first 7 days after surgery
  The VIS will be calculated using the formula:
  Dopamine dose (mcg/Kg/min) + Dobutamine dose (mcg/Kg/min) + 100 x Epinephrine dose (mcg/Kg/min) + 100 x Norepinephrine dose (mcg/Kg/min) + 50 x Levosimendan dose (mcg/Kg/min) + Enoximone dose (mcg/Kg/min) + 10.000 x Vasopressin dose (UI/kg/min).
  The maximum VIS will be recorded each day.
local infections | within 30 days after surgery.
  Postoperative local infections, including pneumonia, deep sternal wound infection/mediastinitis, endocarditis, central line infection, and urinary tract infection.
Other non-cardiac postoperative complications | within 30 days after surgery
  including hepatobiliary disorders, pneumothorax, pleural effusion, and delirium
Quality of life | assessed at 1 year after surgery.
  Quality of life meaurement with the Kansas City Cardiomyopathy Questionnaire (KCCQ) or Activities of Daily Living (ADL) score .
  KCCQ includes 23 items that map to 7 domains: symptom frequency; symptom burden; symptom stability; physical limitations; social limitations; quality of life; and self-efficacy. All scores are represented on a 0-to-100-point scale, where lower scores represent more severe symptoms and/or limitations and scores of 100 indicate no symptoms, no limitations, and excellent quality of life.
  Activities of daily living (ADLs) are important tasks one can do on a regular basis. BasicADLs, incluiding bathing, personal hygiene and grooming, toileting and continence, eating and feeding, dressing, moving/transferring. Katz ADL scale ranges from 0-6, one point for each task can do independently. Higer score stands for more indenpendent in daily life.

CONTACTS AND LOCATIONS:
Overall Officials: Chong Lei, M.D., & phd, Principal Investigator — Xijing Hospital
Locations (3):
- Massachusetts General Hospital, Department of Anesthesia, Critical Care and Pain Medicine, Boston, Massachusetts, United States
- Xijing Hospital, Xi'an, Shaanxi, China
- Cardiology Research Institute, Tomsk National Research Medical Center, Tomsk, Russia

IPD SHARING:
Plan to Share IPD: Yes
The sharing of Individual Patient Data (IPD) will be considered at 1 year after the publication of the primary results of the project. Any request for IPD sharing should be submitted as a proposal to the Principal Investigator (PI), clearly outlining the intended use of the data.
  The Steering Committee of the project will review the proposal and assess whether sharing the data aligns with the project's goals, ethical considerations, and any applicable regulations. Based on this review, the Steering Committee will make a decision regarding the approval of data sharing.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: beginning 12 months after publication of the primary results
Access Criteria: Investigators who provide a methodologically sound proposal and whose proposed use of data has been approved by the steering committee of NORISC. For instance for using IPD data for meta- analysis. Proposals should be submitted to principle investigator and the steering committee of the NORISC trial. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Yan Y, Kamenshchikov N, Zheng Z, Lei C. Inhaled nitric oxide and postoperative outcomes in cardiac surgery with cardiopulmonary bypass: A systematic review and meta-analysis. Nitric Oxide. 2024 May 1;146:64-74. doi: 10.1016/j.niox.2024.03.004. Epub 2024 Mar 29. PMID 38556145
- [Background] Abouzid M, Roshdy Y, Daniel JM, Rzk FM, Ismeal AAA, Hendawy M, Tanashat M, Elnagar M, Daoud N, Ramadan A. The beneficial use of nitric oxide during cardiopulmonary bypass on postoperative outcomes in children and adult patients: a systematic review and meta-analysis of 2897 patients. Eur J Clin Pharmacol. 2023 Nov;79(11):1425-1442. doi: 10.1007/s00228-023-03554-9. Epub 2023 Aug 31. PMID 37650923
- [Background] Strong C, Raposo L, Castro M, Madeira S, Tralhao A, Ventosa A, Rebocho MJ, Almeida M, Aguiar C, Neves JP, Mendes M. Haemodynamic effects and potential clinical implications of inhaled nitric oxide during right heart catheterization in heart transplant candidates. ESC Heart Fail. 2020 Apr;7(2):673-681. doi: 10.1002/ehf2.12639. Epub 2020 Feb 11. PMID 32045139
- [Background] Liu K, Wang H, Yu SJ, Tu GW, Luo Z. Inhaled pulmonary vasodilators: a narrative review. Ann Transl Med. 2021 Apr;9(7):597. doi: 10.21037/atm-20-4895. PMID 33987295
- [Background] Janssens SP, Bogaert J, Zalewski J, Toth A, Adriaenssens T, Belmans A, Bennett J, Claus P, Desmet W, Dubois C, Goetschalckx K, Sinnaeve P, Vandenberghe K, Vermeersch P, Lux A, Szelid Z, Durak M, Lech P, Zmudka K, Pokreisz P, Vranckx P, Merkely B, Bloch KD, Van de Werf F; NOMI investigators. Nitric oxide for inhalation in ST-elevation myocardial infarction (NOMI): a multicentre, double-blind, randomized controlled trial. Eur Heart J. 2018 Aug 1;39(29):2717-2725. doi: 10.1093/eurheartj/ehy232. PMID 29800130
- [Background] Signori D, Magliocca A, Hayashida K, Graw JA, Malhotra R, Bellani G, Berra L, Rezoagli E. Inhaled nitric oxide: role in the pathophysiology of cardio-cerebrovascular and respiratory diseases. Intensive Care Med Exp. 2022 Jun 27;10(1):28. doi: 10.1186/s40635-022-00455-6. PMID 35754072
- [Background] Bowdish ME, D'Agostino RS, Thourani VH, Schwann TA, Krohn C, Desai N, Shahian DM, Fernandez FG, Badhwar V. STS Adult Cardiac Surgery Database: 2021 Update on Outcomes, Quality, and Research. Ann Thorac Surg. 2021 Jun;111(6):1770-1780. doi: 10.1016/j.athoracsur.2021.03.043. Epub 2021 Mar 29. PMID 33794156
- [Background] Schaer DJ, Schaer CA, Humar R, Vallelian F, Henderson R, Tanaka KA, Levy JH, Buehler PW. Navigating Hemolysis and the Renal Implications of Hemoglobin Toxicity in Cardiac Surgery. Anesthesiology. 2024 Dec 1;141(6):1162-1174. doi: 10.1097/ALN.0000000000005109. PMID 39159287
- [Background] Azem K, Novakovsky D, Krasulya B, Fein S, Iluz-Freundlich D, Uhanova J, Kornilov E, Eidelman LA, Kaptzon S, Gorfil D, Aravot D, Barac Y, Aranbitski R. Effect of nitric oxide delivery via cardiopulmonary bypass circuit on postoperative oxygenation in adults undergoing cardiac surgery (NOCARD trial): a randomised controlled trial. Eur J Anaesthesiol. 2024 Sep 1;41(9):677-686. doi: 10.1097/EJA.0000000000002022. Epub 2024 May 28. PMID 39037709
- [Background] Kamenshchikov NO, Anfinogenova YJ, Kozlov BN, Svirko YS, Pekarskiy SE, Evtushenko VV, Lugovsky VA, Shipulin VM, Lomivorotov VV, Podoksenov YK. Nitric oxide delivery during cardiopulmonary bypass reduces acute kidney injury: A randomized trial. J Thorac Cardiovasc Surg. 2022 Apr;163(4):1393-1403.e9. doi: 10.1016/j.jtcvs.2020.03.182. Epub 2020 Jun 25. PMID 32718702
- [Background] Lei C, Berra L, Rezoagli E, Yu B, Dong H, Yu S, Hou L, Chen M, Chen W, Wang H, Zheng Q, Shen J, Jin Z, Chen T, Zhao R, Christie E, Sabbisetti VS, Nordio F, Bonventre JV, Xiong L, Zapol WM. Nitric Oxide Decreases Acute Kidney Injury and Stage 3 Chronic Kidney Disease after Cardiac Surgery. Am J Respir Crit Care Med. 2018 Nov 15;198(10):1279-1287. doi: 10.1164/rccm.201710-2150OC. PMID 29932345
- [Background] Muenster S, Zarragoikoetxea I, Moscatelli A, Balcells J, Gaudard P, Pouard P, Marczin N, Janssens SP. Inhaled NO at a crossroads in cardiac surgery: current need to improve mechanistic understanding, clinical trial design and scientific evidence. Front Cardiovasc Med. 2024 Apr 5;11:1374635. doi: 10.3389/fcvm.2024.1374635. eCollection 2024. PMID 38646153
- [Background] David N, Lakha S, Walsh S, Fried E, DeMaria S Jr. Novel inhaled pulmonary vasodilators in adult cardiac surgery: a scoping review. Can J Anaesth. 2024 Aug;71(8):1154-1162. doi: 10.1007/s12630-024-02770-w. Epub 2024 May 23. PMID 38782851
- [Background] Ghadimi K, Cappiello JL, Wright MC, Levy JH, Bryner BS, DeVore AD, Schroder JN, Patel CB, Rajagopal S, Shah SH, Milano CA; INSPIRE-FLO Investigators. Inhaled Epoprostenol Compared With Nitric Oxide for Right Ventricular Support After Major Cardiac Surgery. Circulation. 2023 Oct 24;148(17):1316-1329. doi: 10.1161/CIRCULATIONAHA.122.062464. Epub 2023 Jul 4. PMID 37401479
- [Background] Benedetto M, Romano R, Baca G, Sarridou D, Fischer A, Simon A, Marczin N. Inhaled nitric oxide in cardiac surgery: Evidence or tradition? Nitric Oxide. 2015 Sep 15;49:67-79. doi: 10.1016/j.niox.2015.06.002. Epub 2015 Jul 14. PMID 26186889